CLINICAL TRIAL: NCT00736840
Title: Pivotal Study to Evaluate the Efficacy and Safety of the BreathID® System for Detection of Cirrhosis Using the ¹³C-methacetin Breath Test(MBT)
Brief Title: BreathID 13C-Methacetin Breath Test for Detecting Cirrhosis
Acronym: MBT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meridian Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: HIS-EX-408
Record Dates: First submitted 2008-08-14; First posted 2008-08-18 (Estimated); Results first posted 2012-03-16 (Estimated); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Chronic Liver Disease
Keywords: Methacetin; Breath; Test; Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CLD (chronic liver disease) (Other): Chronic liver disease subjects with recent biopsy will be tested with a breath tests using a 13C enriched substrate metabolized by their liver
  Interventions: Device: c13 methacetin solution with breath analyzer

INTERVENTIONS:
Device: c13 methacetin solution with breath analyzer — Carbon 13 methacetin 75mg dissolved in 150 ml is given to the subject and metabolism is measured by a breath analyzer after decomposed by the liver

SUMMARY:
This trial is a pivotal trial to validate the use of a 13 C labeled substrate called methacetin and the BreathID automatic breath testing system, for determination of cirrhosis in patients with chronic liver disease.

DETAILED DESCRIPTION:
Patients with chronic liver disease who have a recent biopsy will be offered a breath test. Correlation will be shown between histology and breath test in determining cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 with chronic liver disease

Exclusion Criteria:

* Patients that are taking hepatotoxin drug.
* Patient with severe congestive heart failure
* Patient with severe pulmonary hypertension
* Patient with uncontrolled diabetes mellitus
* Patient with previous surgical bypass surgery for morbid obesity
* Patient with extensive small bowel resection
* Patient currently receiving total parenteral nutrition
* Patient is a recipients of any organ transplant
* Patients that received any anti-viral treatment within the past year
* Women who are pregnant
* Patient allergic to acetaminophen (such as Tylenol or any other related medications)
* Patient with history of chronic obstructive pulmonary disease or symptomatic bronchial asthma
* Patients unable to sign informed consent
* Patients that based on the opinion of the investigator should not be enrolled into this study
* Patients that are participating in other clinical trials evaluating experimental treatments or procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2008-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Gordon, MD, Principal Investigator — Henry Ford Health System; Adrian Rueben, MD, Principal Investigator — Medical University of South Carolina; Gadi Lalazar, MD, Principal Investigator — Hadassah Medical Organization; Arun Sanyal, MD, Principal Investigator — Virginia Commonwealth University; Fred Poordad, MD, Principal Investigator — Cedars Sinai Health System; K Rajender Reddy, MD, Principal Investigator — University of Pennsylvania Health System; Zobair Younossi, MD, Principal Investigator — Inova Health Care Services; Arthur McCullough, MD, Principal Investigator — The Cleveland Clinic; John Vierling, MD, Principal Investigator — St. Luke's Episcopal Hospital, Baylor College of Medicine; Alexander Fich, MD, Principal Investigator — Soroka University Medical Center; Eli Zuckerman, MD, Principal Investigator — Carmel Medical Center
Locations (11):
- United States (8):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Henry Ford Health Sytem, Detroit, Michigan
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - St Luke's Episcopal Hospital, Baylor College of Medicine, Houston, Texas
  - Inova Helath System, Falls Church, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
- Israel (3):
  - Soroka Medical Center, Beersheba
  - Carmel Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 414 subjects were collected in 11 sites; 8 in the United states and 3 in Israel. Recruitment began in August 2008 and was completed Sep 2009.
Pre-assignment Details: 4 sites, 1 in Israel and 3 in the United States recruited most of the subjects. Patients with chronic liver disease and recent biopsies performed or planned were approached. Exclusion criteria focused mostly on issues that would affect accuracy of breath test.
Groups:
- CLD (Chronic Liver Disease): Chronic liver disease subjects with recent (within 3 months)liver biopsy will be tested with the 13C methacetin breath test, which entails connecting the subject via a nasal cannula to the BreathID analyzer and after measuring baseline breath, have the subject drink 150cc of aqueous solution which contains 75 mg of 13C -labeled methacetin (Intervention material)
Period: Overall Study
Arm/Group | CLD (Chronic Liver Disease)
Started | 414
Completed | 401 (9 subjects-no biopsy results, 2-no breath test, 2 no biopsy results and no complete breath test)
Not Completed | 13
Not completed — Lost to Follow-up | 13

BASELINE CHARACTERISTICS:
Arm/Group | CLD (Chronic Liver Disease)
Number analyzed (Participants) | 414
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 374
  >=65 years | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178
  Male | 236
Region of Enrollment [Number; unit: participants]
  United States | 327
  Israel | 87

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Likelihood of Cirrhosis Based on "Hepatic Impairment Score" (HIS)
Description: "Hepatic Impairment Score" (HIS) is a score based on breath test parameters and demographic parameters of the subject being tested. A HIS value greater than 0.14 would mean that the subject is likely to be cirrhotic (based on biopsy result as the gold standard). The HIS is a probability score,i.e. ranges from 0 to 1, where 0 would mean the lowest probability of having liver cirrhosis and 1 would be the highest probability of having liver cirrhosis. This would be compared to the actual biopsy result of cirrhosis detection as the gold standard.
Time Frame: Study day 1 after a 1 hour test
Population: The primary efficacy was conducted on all evaluable subject data in the full analysis (FA)set with biopsy confirmed cirrhosis.
Measure: Number; unit: Participants
Arm/Group | CLD (Chronic Liver Disease)
Number analyzed (Participants) | 146
Participants | 146 [66.07 to 80.88]
Statistical Analysis 1: Comparison: CLD (Chronic Liver Disease); The null hypothesis was sensitivity lower than 0.8. We assumed a sensitivity of 0.89 and required a power of 90% to test the hypothesis at a 5% level of significance, and calculated that 173 cirrhotic and 241 non-cirrhotic subjects were needed (for a one-sample binomial test of outcome versus constant); Test type: Non-Inferiority or Equivalence — Provided above; p = 0.0924, Exact binomial test; Sensitivity = 0.74, 95% CI 2-sided [0.6607 to 0.8809], Standard Error of Mean 0.0363

2. Secondary Outcome: AUC of ROC (Area Under Receiver Operating Characteristic Curve)
Description: The AUC represents a summary measure of the ROC curve and is the accuracy of the HIS in detecting cirrhosis compared to the gold standard of biopsy.
Time Frame: At study day 1 after 1 hour test
Measure: Mean (95% Confidence Interval); unit: Probability
Arm/Group | CLD (Chronic Liver Disease)
Number analyzed (Participants) | 414
Probability | 0.785 [0.737 to 0.834]
Statistical Analysis 1: Comparison: CLD (Chronic Liver Disease); Test type: Non-Inferiority or Equivalence — Sample size was calculated to enable the testing of both study hypotheses (together) with at least 80% power. Our best estimate of sensitivity of the HIS diagnosis in the population, was 0.9 and its specificity 0.79. Requiring a power of 90% for each of the hypotheses and a 5% level of significance, to test the null hypotheses 173 cirrhotic and 241 non-cirrhotic subjects were needed.Therefore a total of at least 414 subjects were required; p < 0.0001, Regression, Logistic; AUC ROC = 0.785, 95% CI 2-sided [0.737 to 0.834], Standard Error of Mean 0.0485

ADVERSE EVENTS:
Arm/Group | CLD (Chronic Liver Disease)
Serious Adverse Events (participants affected / at risk) | 0/414
Other Adverse Events (participants affected / at risk) | 0/414

LIMITATIONS AND CAVEATS:
Technical problems caused the termination of 2 subjects who did not complete breath test. Liver biopsy, 1 patient refused and others had signs of HCC thus disqualified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any manuscript, abstract or other publication or presentation of results or information arising from the study (including ancillary studies involving trial patients) must be prepared in conjunction with Exalenz. Such materials must be submitted to Exalenz for review and comment at least 30 days prior to submission for publication or presentation.